CLINICAL TRIAL: NCT04754451
Title: The Efficacy and Safety of 5% Lidocaine Patch for Postoperative Pain in Unilateral Inguinal Herniorrhaphy
Brief Title: The Effect of Lidocaine Patch for Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BON WOOK KOO (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, BON WOOK KOO, associative professor of anesthesiology, Seoul National University Bundang Hospital
Organization: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDPS
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P(placebo) (No Intervention): Attach two placebo patches for 12 hours, above and below the incision site.
- Group L(lidocaine patch) (Experimental): Attach two lidocaine patches for 12 hours, above and below the incision site.
  Interventions: Drug: Group L

INTERVENTIONS:
Drug: Group L — Attach two lidocaine patches for 12 hours, one above and below the incision site.
  Other Names: lidotopcaplasma
  Arms: Group L(lidocaine patch)

SUMMARY:
The lidocaine patch is currently only permitted for post herpetic neuralgia but the investigators want to study its effectiveness in post operative pain after inguinal herniorrhaphy

DETAILED DESCRIPTION:
After open unilateral inguinal herniorrhaphy, patients are randomly divided into group L and group P groups. Group L attaches two lidocaine patches for 12 hours, above and below the incision site. Group P attaches two placebo patches for 12 hours, above and below the incision site. Pain scores are recorded for 30 minutes, 2 hours, 24 hours, and 1 week after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I - II
* Scheduled open unilateral herniorrhaphy

Exclusion Criteria:

* body mass index (BMI) < 18.5 or ≥ 35 kg/m2
* severe renal or hepatic dysfunction
* allergy to amide-based local anesthetic agents
* taking class 1 antiarrhythmic drugs (tocainide and mexiletine, etc.)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The pain score | 24 hours after the anesthesia finished.
  VAS(visual analog scale) measurement for 24 hours after surgery(0-10) 0: no pain 10: severe pain

SECONDARY OUTCOMES:
The pain score | 30 min after the anesthesia finished.
  VAS(visual analog scale) measurement for 24 hours after surgery(0-10) 0: no pain 10: severe pain
The pain score | 2 hours after the anesthesia finished.
  VAS(visual analog scale) measurement for 24 hours after surgery(0-10) 0: no pain 10: severe pain
Total amount of cumulative analgesics | 24 hours after the anesthesia finished.
  total amount of analgesics are measured for 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: BON WOOK KOO, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Universuty, Bundang Hospital, Seongnam-si, Gyonggido, South Korea

REFERENCES:
- [Derived] Ahn HM, Oh HK, Kim DW, Kang SB, Koo BW, Lee PB. Efficacy and safety of 5% lidocaine patches for postoperative pain management in patients undergoing unilateral inguinal hernia repair: study protocol for a prospective, double-blind, randomized, controlled clinical trial. Trials. 2022 Sep 11;23(1):767. doi: 10.1186/s13063-022-06700-3. PMID 36089597